CLINICAL TRIAL: NCT00489411
Title: A Phase III Double Blind Trial of Oral Duloxetine for Treatment of Pain Associated With Chemotherapy-Induced Peripheral Neuropathy
Brief Title: Duloxetine in Treating Peripheral Neuropathy Caused by Chemotherapy in Patients With Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: CALGB-170601; CALGB-170601; CDR0000553389 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Neurotoxicity; Pain; Peripheral Neuropathy; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; neurotoxicity; pain; peripheral neuropathy
MeSH Terms: conditions — Neurotoxicity Syndromes; Pain; Peripheral Nervous System Diseases | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I/Group A (Duloxetine then Placebo) (Experimental): Patients receive oral duloxetine hydrochloride once or twice daily in weeks 1-6. After a 1-week rest period, patients cross over to receive an oral placebo once or twice daily in weeks 8-13.
  Interventions: Drug: duloxetine hydrochloride; Other: placebo
- Arm II/Group B (Placebo then Duloxetine) (Experimental): Patients receive an oral placebo once or twice daily in weeks 1-6. After a 1-week rest period, patients cross over to receive oral duloxetine hydrochloride once or twice daily in weeks 8-13.
  Interventions: Drug: duloxetine hydrochloride; Other: placebo

INTERVENTIONS:
Drug: duloxetine hydrochloride — Given orally
Other: placebo — Given orally

SUMMARY:
RATIONALE: Duloxetine may lessen peripheral neuropathy caused by chemotherapy. It is not yet known whether duloxetine is more effective than a placebo in treating peripheral neuropathy caused by chemotherapy.

PURPOSE: This randomized phase III trial is studying duloxetine to see how well it works compared with a placebo in treating peripheral neuropathy caused by chemotherapy in patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of duloxetine hydrochloride in cancer patients with painful chemotherapy-induced (taxane or platinum agent) peripheral neuropathy.

Secondary

* Determine the influence of this drug on peripheral neuropathy-related functional status and quality of life of these patients.
* Describe the differences in duloxetine hydrochloride efficacy when used to treat pain caused by chemotherapy-induced peripheral neuropathy based on the neurotoxic drug and class.

OUTLINE: This is a randomized, double-blind, placebo-controlled, crossover study. Patients are stratified according to prior neurotoxic agent (paclitaxel vs oxaliplatin vs other taxane agents without paclitaxel vs platinum agents [cisplatin] without oxaliplatin) and high risk for developing painful chemotherapy-induced peripheral neuropathy (no vs yes). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral duloxetine hydrochloride once or twice daily in weeks 1-6. After a 1-week rest period, patients cross over to receive an oral placebo once or twice daily in weeks 8-13.
* Arm II: Patients receive an oral placebo once or twice daily in weeks 1-6. After a 1-week rest period, patients cross over to receive oral duloxetine hydrochloride once or twice daily in weeks 8-13.

Patients complete pain and quality of life questionnaires, including the BPI-SF once weekly and FACT/GOG-NTX and EORTC QLQ-C30 questionnaires, in weeks 1, 6, 8, and 13.

After completion of study treatment, patients are followed for 2 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer

  * CNS malignancy allowed with the exception of leptomeningeal carcinomatosis
* Must have painful sensory chemotherapy-induced peripheral neuropathy (CIPN) resulting from prior treatment with single-agent taxane or platinum agents (paclitaxel, docetaxel, nab-paclitaxel, oxaliplatin, cisplatin) (may not have received drugs from both classes)

  * CIPN > grade 1 as measured by NCI-CTCAE v 4.0
  * Average neuropathic pain score ≥ 4
* Patients with the following illnesses known to cause peripheral neuropathy are eligible, provided they have no evidence of neuropathy from these illnesses:

  * Diabetes mellitus
  * Peripheral vascular disease
  * HIV infection
  * Significant degenerative or familial neurologic disorder known to cause peripheral neuropathy
* No clinical or subclinical neuropathy from nerve compression injuries (i.e., carpal tunnel syndrome, brachial plexopathy, spinal stenosis, or spinal nerve root compression)

PATIENT CHARACTERISTICS:

* AST ≤ 3 times upper limit of normal
* Total bilirubin ≤ normal
* Creatinine clearance > 30 mL/min
* Not pregnant or nursing
* Able to take oral or enteral medication
* No history of seizure disorder
* No diagnosis of ethanol addiction or dependence within the past 10 years
* No history of narrow-angle glaucoma
* None of the following:

  * History of suicidal thoughts
  * Symptoms of or history of schizophrenia, bipolar disease, or a major depression
  * Serious eating disorder such as bulimia or anorexia where electrolyte imbalance is likely

PRIOR CONCURRENT THERAPY:

* At least 3 months since prior and no concurrent taxane or platinum agent
* At least 14 days since prior and no concurrent monoamine oxidase inhibitors or other antidepressants
* No other prior or concurrent neurotoxic drugs (e.g., vincristine, vinblastine, cytarabine, thalidomide, bortezomib, carboplatin, or procarbazine)
* No concurrent anticonvulsants
* No concurrent B or E vitamin supplementation in doses greater than the recommended daily allowance (RDA)

  * Centrum (standard formula) and One-A-Day "essential" formula which contain 100% RDA for vitamins B6, E, and B12 allowed
  * Other multivitamins allowed provided they contain no more than 100% RDA of B vitamins and vitamin E
* No concurrent treatment (pharmacologic) for depression

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2008-04; Primary Completion 2012-01 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen L. Smith, PhD, ARNP, AOCN, Study Chair — University of Michigan
Locations (475):
- United States (475):
  - Kaiser Permanente - Deer Valley, Antioch, California
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Cancer Care Center at John Muir Health - Concord Campus, Concord, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Valley Medical Oncology, Fremont, California
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Camino Medical Group - Treatment Center, Mountain View, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Kaiser Permanente - Division of Research - Oakland, Oakland, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - Pismo Beach, California
  - Kaiser Permanente Medical Center - Rancho Cordova, Rancho Cardova, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Sutter Health - Western Division Cancer Research Group, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Sutter Solano Medical Center, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Kaiser Permanente - Denver, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente - Lafayette, Lafayette, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Bendheim Cancer Center at Greenwich Hospital, Greenwich, Connecticut
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Kaiser Permanente - Moanalua Medical Center and Clinic, Honolulu, Hawaii
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Central Dupage Cancer Center, Warrenville, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Cancer Resource Center at King's Daughters Medical Center, Ashland, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Shore Regional Cancer Center at Memorial Hospital - Easton, Easton, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton MD, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Great Lakes Cancer Institute at McLaren Regional Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Michiana Hematology Oncology PC - Niles, Niles, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls Medical Group, PA, Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - St. Anthony's Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - Comprehensive Cancer Care, PC, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center at Catholic Medical Center, Manchester, New Hampshire
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - New York Oncology Hematology, PC at Albany Regional Cancer Care, Albany, New York
  - New York Oncology Hematology, PC at Albany Medical Center, Albany, New York
  - Amsterdam Community Cancer Program, Amsterdam, New York
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - New York Oncology Hematology, PC - Hudson, Hudson, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - New York Oncology Hematology, PC - Latham, Latham, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Riverview Cancer Care Medical Associates, PC, Rexford, New York
  - Nalitt Cancer Institute at Staten Island University Hospital, Staten Island, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Samaritan Hospital at Northeast Health, Troy, New York
  - Dickstein Cancer Treatment Center at White Plains Hospital Center, White Plains, New York
  - Waverly Hematology Oncology, Cary, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - CaroMont Cancer Center at Gaston Memorial Hospital, Gastonia, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Emerywood Hematology/Oncology, High Point, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Trinity CancerCare Center, Minot, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Bay Area Hospital, Coos Bay, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Doylestown Hospital Cancer Center, Doylestown, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Cancer Center at Phoenixville Hospital, Phoenixville, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Self Regional Cancer Center at Self Regional Medical Center, Greenwood, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Martha Jefferson Hospital Cancer Care Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - Aurora Memorial Hospital of Burlington, Burlington, Wisconsin
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Vince Lombardi Cancer Center at Aurora Lakeland Medical Center - Elkhorn, Elkhorn, Wisconsin
  - Oncology Alliance - Franklin, Franklin, Wisconsin
  - Oncology Alliance, SC - Milwaukee - East, Glendale, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercy Regional Cancer Center, Janesville, Wisconsin
  - Oncology Alliance - Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic - Marinette, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Aurora Advanced Healthcare East Mequon Clinic, Mequon, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Medical Consultants, Limited, Milwaukee, Wisconsin
  - Oncology Alliance, SC - Milwaukee - South, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Health Center - Racine, Racine, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic - Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic - Two Rivers, Two Rivers, Wisconsin
  - Aurora Health Center - Waukesha, Waukesha, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Oncology Alliance, SC - Milwaukee - West, Wauwatosa, Wisconsin
  - Aurora Women's Pavilion of West Allis Memorial Hospital, West Allis, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Lavoie Smith EM, Pang H, Cirrincione C, et al.: CALGB 170601: A phase III double blind trial of duloxetine to treat painful chemotherapy-induced peripheral neuropathy (CIPN). [Abstract] J Clin Oncol 30 (Suppl 15): A-CRA9013, 2012.
- [Derived] Smith EM, Pang H, Ye C, Cirrincione C, Fleishman S, Paskett ED, Ahles T, Bressler LR, Le-Lindqwister N, Fadul CE, Loprinzi C, Shapiro CL; Alliance for Clinical Trials in Oncology. Predictors of duloxetine response in patients with oxaliplatin-induced painful chemotherapy-induced peripheral neuropathy (CIPN): a secondary analysis of randomised controlled trial - CALGB/alliance 170601. Eur J Cancer Care (Engl). 2017 Mar;26(2):10.1111/ecc.12421. doi: 10.1111/ecc.12421. Epub 2015 Nov 25. PMID 26603828
- [Derived] Smith EM, Pang H, Cirrincione C, Fleishman S, Paskett ED, Ahles T, Bressler LR, Fadul CE, Knox C, Le-Lindqwister N, Gilman PB, Shapiro CL; Alliance for Clinical Trials in Oncology. Effect of duloxetine on pain, function, and quality of life among patients with chemotherapy-induced painful peripheral neuropathy: a randomized clinical trial. JAMA. 2013 Apr 3;309(13):1359-67. doi: 10.1001/jama.2013.2813. PMID 23549581

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of screened and the number offered participation but declined was not captured.
Groups:
- Arm I/Group A (Duloxetine Then Placebo): Patients will take one capsule of 30 mg duloxetine orally daily for 7 days (week 1), and then increase to two capsules of duloxetine (60 mg duloxetine) orally daily for 28 days (weeks 2-5). Duloxetine will be tapered during week 6 (one capsule daily for 7 days), and will be discontinued during week 7 (no capsules for 7 days). Patients will then cross over to receive the alternative treatment (placebo), and the sequence will be repeated. Patients will take one capsule of placebo daily for 7 days (week 8), two capsules of placebo daily for 28 days (weeks 9-12), one capsule of placebo daily for 7 days (week 13), and then no capsules for 7 days (week 14).
- Arm II/Group B (Placebo Then Duloxetine): Patients will take one capsule of placebo orally daily for 7 days (week 1), and then increase to two capsules of placebo orally daily for 28 days (weeks 2-5). Placebo will be tapered during week 6 (one capsule daily for 7 days), and will be discontinued during week 7 (no capsules for 7 days). Patients will then cross over to receive the alternative treatment (duloxetine), and the sequence will be repeated. Patients will take one capsule of duloxetine daily for 7 days (week 8), two capsules of duloxetine daily for 28 days (weeks 9-12), one capsule of duloxetine daily for 7 days (week 13), and then no capsules for 7 days (week 14).
Period: Initial Treatment Period (Weeks 1-5)
Arm/Group | Arm I/Group A (Duloxetine Then Placebo) | Arm II/Group B (Placebo Then Duloxetine)
Started | 115 | 116
Completed | 87 | 94
Not Completed | 28 | 22
Not completed — Withdrew consent prior to intervention | 6 | 5
Not completed — Discontinued study drug early | 21 | 12
Not completed — Incomplete data | 1 | 5
Period: Washout Period (Weeks 6-7)
Arm/Group | Arm I/Group A (Duloxetine Then Placebo) | Arm II/Group B (Placebo Then Duloxetine)
Started | 87 | 94
Completed (Reasons for why patients did not participate in the crossover treatment period were not captured.) | 85 | 93
Not Completed | 2 | 1
Period: Crossover Treatment Period (Weeks 8-12)
Arm/Group | Arm I/Group A (Duloxetine Then Placebo) | Arm II/Group B (Placebo Then Duloxetine)
Started | 85 | 93
Completed | 67 | 74
Not Completed | 18 | 19
Not completed — Discontinued intervention early | 11 | 12
Not completed — Incomplete data | 7 | 7

BASELINE CHARACTERISTICS:
Population: All patients who received duloxetine/placebo as randomized were included in the analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I/Group A (Duloxetine Then Placebo) | Arm II/Group B (Placebo Then Duloxetine) | Total
Number analyzed (Participants) | 109 | 111 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (10.4) | 59.0 (10.6) | 59.0 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 67 | 138
  Male | 38 | 44 | 82
Region of Enrollment [Number; unit: participants]
  United States | 109 | 111 | 220

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Pain From Week 1 to Week 5, as Measured by the BPI-SF Average Pain Severity Item
Description: Change in average pain from Week 1 to Week 5, measured on day 1 of Weeks 1 and 6 by the Brief Pain Inventory Short Form (BPI-SF) was calculated as value at Day 1 of Week 1 minus value at Day 1 of Week 6 to yield positive improvement values. The BPI-SF contains 4 items assessing average, worst, least, and intermediate pain severity in the last 24 hours. Pain severity items are scored using an 11-point numeric rating scale (0, no pain; 10, pain as bad as you can imagine). Average pain severity was chosen as the primary outcome based on recommendations from the Initiative on Methods, Measurements, and Pain Assessment in Clinical Trials (IMMPACT). Patients completed the BPI-SF when thinking only about pain from peripheral neuropathy. The Cronbach's alpha reliability for the BPI ranges between 0.77 and 0.91. The comparison of interest was the difference between the 2 treatment groups in pain change during the initial treatment period.
Time Frame: Day 1 of Week 1 to Day 1 of Week 6
Population: Patients who completed initial intervention (prior to crossing over to receive alternate study drug duloxetine or placebo) and had complete data were included in the primary analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm I/Group A (Duloxetine Then Placebo) | Arm II/Group B (Placebo Then Duloxetine)
Number analyzed (Participants) | 87 | 94
units on a scale | 1.06 [0.72 to 1.40] | 0.34 [0.01 to 0.66]
Statistical Analysis 1: Comparison: Arm I/Group A (Duloxetine Then Placebo) vs Arm II/Group B (Placebo Then Duloxetine); Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney); Mean Difference = 0.73, 95% CI 2-sided [0.26 to 1.20]

2. Secondary Outcome: Change in Pain-related Functional Interference Score From Week 1 to Week 5, as Measured by the BPI-SF Interference Score
Description: Change in pain-related functional interference score during the initial treatment period (Week 1 to Week 5), as measured by the BPI-SF interference score: Using an accepted method for accessing the influence of pain on function, 7 BPI-SF items were used to quantify the degree to which pain interfered with daily activities or function (0, does not interfere; 10 completely interferes). The 7 items were summed to obtain a total interference score, which ranged from 0 to 70, with lower scores meaning less interference. The mean change in pain-related functional interference score during the initial treatment period are reported below for each treatment arm and was calculated as value at Day 1 of Week 1 minus value at Day 1 of Week 6 to yield positive improvement values.
Time Frame: Day 1 of Week 1 to Day 1 to Week 6
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm I/Group A (Duloxetine Then Placebo) | Arm II/Group B (Placebo Then Duloxetine)
Number analyzed (Participants) | 87 | 94
units on a scale | 7.9 [5.4 to 10.5] | 3.5 [1.1 to 5.9]
Statistical Analysis 1: Comparison: Arm I/Group A (Duloxetine Then Placebo) vs Arm II/Group B (Placebo Then Duloxetine); Test type: Superiority or Other; Mean Difference = 4.40, 95% CI 2-sided [0.93 to 7.88]

3. Secondary Outcome: Change in the Total Score of the FACT/COG-NTX From Week 1 to Week 5
Description: Patient-reported QOL was assessed using the Functional Assessment of Cancer Treatment, Gynecologic Oncology Group Neurotoxicity (FACT/GOG-Ntx) subscale on day 1 of weeks 1, 6, 8, and 13. The instrument contains 11 questions, assessing numbness, tingling, and discomfort in the hands or feet; difficulty hearing; tinnitus; joint pain or muscle cramps; weakness; or trouble walking, buttoning buttons, or feeling small shapes when placed in the hand. Items are scored from 0 to 4 (o, not at all; 4, very much) and summed (total score range, 0-44, with higher scores indicating a worse outcome). A 2- to 3-point change is defined as a clinically meaningful improvement in QOL per published recommendations specific to similar measures. The Mean Change During Initial Treatment Period in the FACT/GOG-Ntx total score are reported for each treatment arm and was calculated as value at Day 1 of Week 1 minus value at Day 1 of Week 6 to yield positive improvement values.
Time Frame: Day 1 of Week 1 to Day 1 of Week 6
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm I/Group A (Duloxetine Then Placebo) | Arm II/Group B (Placebo Then Duloxetine)
Number analyzed (Participants) | 87 | 94
units on a scale | 2.44 [0.43 to 4.45] | 0.87 [-1.09 to 2.82]
Statistical Analysis 1: Comparison: Arm I/Group A (Duloxetine Then Placebo) vs Arm II/Group B (Placebo Then Duloxetine); Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney); Mean Difference = 1.58, 95% CI 2-sided [0.15 to 3.00]

4. Secondary Outcome: Change in Average Pain From Week 8 to Week 12, as Measured by the BPI-SF Average Pain Severity Item
Description: Change in average pain from Week 8 to Week 12, measured on day 1 of Weeks 8 and 13 by the Brief Pain Inventory Short Form (BPI-SF) was calculated as value at Day 1 of Week 8 minus value at Day 1 of Week 13 to yield positive improvement values. The BPI-SF contains 4 items assessing average, worst, least, and intermediate pain severity in the last 24 hours. Pain severity items are scored using an 11-point numeric rating scale (0, no pain; 10, pain as bad as you can imagine). Average pain severity was chosen as the primary outcome based on recommendations from the Initiative on Methods, Measurements, and Pain Assessment in Clinical Trials (IMMPACT). Patients completed the BPI-SF when thinking only about pain from peripheral neuropathy. The Cronbach's alpha reliability for the BPI ranges between 0.77 and 0.91. The comparison of interest was the difference between the 2 treatment groups in pain change during the crossover treatment period.
Time Frame: Day 1 of Week 8 to Day 1 of Week 13
Population: Patients who completed crossover intervention and had complete data were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm I/Group A (Duloxetine Then Placebo) | Arm II/Group B (Placebo Then Duloxetine)
Number analyzed (Participants) | 67 | 74
units on a scale | 0.41 [0.06 to 0.89] | 1.42 [0.97 to 1.87]
Statistical Analysis 1: Comparison: Arm I/Group A (Duloxetine Then Placebo) vs Arm II/Group B (Placebo Then Duloxetine); Test type: Superiority or Other; Mean difference = 1.01, 95% CI 2-sided [0.36 to 1.65]

ADVERSE EVENTS:
Time Frame: Adverse events are assessed during weeks 1-15 of the study.
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. All graded adverse events are reported. AEs are presented "per sequence" based on how they were collected in the study. The Number of Participants at Risk include subjects who received an intervention, did not have incomplete AE data during primary analysis, and did not withdraw consent prior to receiving the intervention.
Arm/Group | Arm I/Group A (Duloxetine Then Placebo) | Arm II/Group B (Placebo Then Duloxetine)
Serious Adverse Events (participants affected / at risk) | 1/108 | 3/107
Other Adverse Events (participants affected / at risk) | 93/108 | 91/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I/Group A (Duloxetine Then Placebo) (N=108) | Arm II/Group B (Placebo Then Duloxetine) (N=107)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I/Group A (Duloxetine Then Placebo) (N=108) | Arm II/Group B (Placebo Then Duloxetine) (N=107)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 1 (4)
Vision blurred (Eye disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 29 (84) | 32 (96)
Diarrhea (Gastrointestinal disorders) | 28 (59) | 31 (103)
Dry mouth (Gastrointestinal disorders) | 24 (116) | 27 (146)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (7)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (4)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 50 (88) | 40 (82)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 1 (3)
Vomiting (Gastrointestinal disorders) | 6 (6) | 4 (4)
Chest pain (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 2 (6) | 1 (2)
Fatigue (General disorders) | 56 (205) | 50 (297)
Fever (General disorders) | 0 (0) | 1 (1)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (9) | 3 (11)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 2 (4) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (2) | 1 (1)
Serum cholesterol increased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 16 (26) | 23 (83)
Blood glucose increased (Metabolism and nutrition disorders) | 4 (7) | 2 (16)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (30)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (20) | 7 (58)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 12 (33) | 23 (69)
Dizziness (Nervous system disorders) | 24 (56) | 19 (49)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (5)
Headache (Nervous system disorders) | 29 (74) | 28 (97)
Memory impairment (Nervous system disorders) | 1 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 5 (22) | 3 (17)
Peripheral motor neuropathy (Nervous system disorders) | 3 (14) | 3 (26)
Peripheral sensory neuropathy (Nervous system disorders) | 21 (166) | 26 (205)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (2)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 39 (167) | 40 (223)
Glomerular filtration rate decreased (Renal and urinary disorders) | 2 (5) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Ejaculation disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (5)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 4 (13) | 4 (23)
Hypertension (Vascular disorders) | 2 (2) | 3 (7)
Hypotension (Vascular disorders) | 0 (0) | 1 (2)
Vascular disorder (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes